CLINICAL TRIAL: NCT02768506
Title: Non-randomized Prospective Comparison Between SADI-S and Gastric Bypass for the Treatment of Morbid Obesity and Its Associated Co-morbidities
Brief Title: Prospective Comparison Between SADI-S and Gastric Bypass
Acronym: SADI-S-GB
Status: Completed | Type: Observational
Sponsor: Hospital San Carlos, Madrid (Other)
Responsible Party: Principal Investigator, Andres Sanchez-Pernaute, PhD, MD, Hospital San Carlos, Madrid
Other Study IDs: ASP-004
Record Dates: First submitted 2016-05-08; First posted 2016-05-11 (Estimated); Last update posted 2016-05-11 (Estimated); Status verified 2016-05

CONDITIONS: Morbid Obesity; Diabetes
Keywords: obesity, malabsorption, gastric bypass, SADI-S
MeSH Terms: conditions — Obesity, Morbid; Diabetes Mellitus; Obesity; Malabsorption Syndromes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Liver biopsy
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Gastric bypass: Subjects submitted to gastric bypass
- SADI-S: Subjects submitted to SADI-S

SUMMARY:
Patients with BMI over 40 or with BMI over 35 and comorbidities are offered SADI-S with a variable limb length between 250 cm and 300 cm or gastric bypass.

Results on weight loss, comorbidities resolution, complications, re-operations, need of supplements are registered.

DETAILED DESCRIPTION:
Morbid obese patients and patients with an initial BMI over 35 with associated comorbidities - as diabetes mellitus - are evaluated for bariatric surgery. Candidates are offered a standard gastric bypass or a single anastomosis duodeno-ileal bypass with sleeve gastrectomy. Patients with higher BMI and those with worse metabolic condition are encouraged to accept the malabsorptive option.

Gastric bypass is performed with a 150 cm alimentary limb and a calibrated pouch and anastomosis over a 14 mm bougie. SADI-S is performed with a sleeve gastrectomy over a 54 French (18 mm) gastric bougie and a 250 cm common limb.

Patients are managed equally during admission: 6 hours to initiate oral intake, 2 days to remove abdominal drain and 3 days to discharge unless contraindicated. Follow up is performed through visits every 3 months the first 2 postoperative years and every 6 months from the 3rd to the 5th year.

ELIGIBILITY:
Inclusion Criteria:

* Morbid obesity

Exclusion Criteria:

* Drug addiction
* Alcoholic
* Neoplasms
* Immunosuppression
* Mental diseases

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Morbid obesity patients asking for surgery
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2009-09; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Weight loss | 5 years
  Excess weight loss percentage and total weight loss percentage in the first 5 years

SECONDARY OUTCOMES:
Diabetes remission | 5 years
  Normalization of glycemia and HbA1c with no anti-diabetic medications

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Clínico San Carlos, Madrid, Madrid, Spain